CLINICAL TRIAL: NCT02033226
Title: Evaluation of Clinical, Anti-Inflammatory and Anti-Infective Properties of Amniotic Membranes Used For Guided Tissue Regeneration in Contained Defects
Brief Title: Clinical, Anti-Inflammatory And Anti-Infective Properties Of Amniotic Membranes Used For Guided Tissue Regeneration
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SVS Institute of Dental Sciences (Other)
Responsible Party: Principal Investigator, Dr R Viswa Chandra, Primary Investigator and Director of Records, SVS Institute of Dental Sciences
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: SVS031101
Record Dates: First submitted 2014-01-08; First posted 2014-01-10 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Chronic Periodontitis
Keywords: Periodontitis; Periodontal Regeneration; Amniotic membrane; Guided tissue regeneration; Anti-inflammatory; Periodontal Therapy.
MeSH Terms: conditions — Chronic Periodontitis; Periodontitis | interventions — Biological Dressings; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amniotic Membrane (Experimental): The test site was treated as follows; After placement and proper condensation of natural Hydroxyapatite graft in the defect, AM was cut based on defect anatomy of surgical site and then adapted over the bone graft and alveolar bone extending from base of the flap reflection to the tooth surface.
  Interventions: Device: Amniotic Membrane
- Control group (Hydroxyapatite only) (Placebo Comparator): The control site was treated by graft placement (Hydroxyapatite) only
  Interventions: Device: Control group (Hydroxyapatite only)

INTERVENTIONS:
Device: Amniotic Membrane — AM strongly resembles the oral mucosal basement membrane and possesses several types of laminins, which can promote regeneration, accelerate tissue adhesion, and preserve tissues, all of which play a key role in improved healing of periodontal lesions and might result in reduction in probing pocket depth (PPD) and decrease in clinical attachment loss (CAL)
  Other Names: TMH Tissue Bank, Mumbai, India
  Arms: Amniotic Membrane
Device: Control group (Hydroxyapatite only) — The placebo group was treated with Hydroxyapatite graft placement only.
  Arms: Control group (Hydroxyapatite only)

SUMMARY:
The objective of this study is to evaluate the anti-inflammatory and anti-infective properties of amniotic membrane (AM) when used for guided tissue regeneration (GTR) in periodontal bone defects.

DETAILED DESCRIPTION:
Study design including Randomization and Blinding The study was designed as a split-mouth, double-blind, randomized controlled clinical trial. Randomization and blinding included computerized generation of the allocation sequence in random permuted blocks (block randomization) and blinded disbursement of medication. Allocation was performed by assigning the block of sites to study groups according to the specified sequence. Based on the sequence, the first operator selected two sites for each of the following experimental sites; the test site, in which amniotic membrane with the graft was placed and the control site which was treated by graft placement only. All the surgeries were performed by a designated operator for the sake of uniformity whereas the relevant readings were recorded by the first operator who was blinded to the nature of the site. The blind was not broken until this clinical trial was completely finished.

After the prospective interdental areas were probed buccally and lingually/palatally, the site was considered for the study if the average probing pocket depth (PPD) was ≥5 mm. All baseline (on the day of surgery) values were recorded before the surgical procedure. Gingival crevicular fluid (GCF) samples for IL-1β were taken at baseline and 1 week and for hBD-2 were taken at baseline, 1 week and 4 weeks. Non-invasive site-specific measures of the plaque index (PI) and modified gingival index (MGI) at the baseline, 1 week, 12 weeks and 24 weeks. The PPD, CAL and bone fill were recorded at the baseline (on the day of surgery) and at the end of 12 and 24 weeks. PPD and CAL were recorded at the baseline and at the end of 12 and 24 weeks using a UNC-15 color-coded periodontal probe. A custom acrylic stent limited to the occlusal 2/3rds of the clinical crown was prepared from a cast obtained from an alginate impression. A groove was prepared in the stent to standardize the probing angulation throughout the procedure and also during the follow up visits.

Radiograph Standardization Standard digital radiographs were taken at baseline, 12 and 24 weeks by the paralleling/long-cone technique at pre-set parameters using a commercially available RVG system. After the imaging plate was placed in the film holder for paralleling technique, addition silicon impression material was added around the biting surface and allowed to set. This arrangement ensured standardized alignment of the aiming device and the holder ensuring correct positioning of the collimator in subsequent radiographs.

Collection of GCF Samples:

After isolation, 6 mm diameter filter paper circles were used for collecting the samples by the intra-crevicular method. The fluid seeping out of the sulcus was collected and any paper contaminated with blood or saliva was discarded, and the collection was repeated after 30 minutes. GCF samples were eluted from the strips by placing them in Eppendorf tubes that contained 500 µL of buffer and stored at -80ºC. GCF Samples were collected at baseline, at the end of 1 and 4 weeks.

Enzyme Linked Immunosorbent Assay (ELISA) for IL-1ß and hBD-2 Commercially available ELISA kits were used to quantify GCF levels of IL-1ß and hBD-2. All assay procedures were conducted according to the manufacturer's instructions and in both the tests, 100μl of the samples or standards were added into the respective wells in duplicate. Color development was stopped using 1% H2SO4 and absorbance of the entire plate was measured within 30 minutes by an ELISA reader at 450nm. The amounts of IL-1ß and hBD-2 were calculated based on the dilutions, and the results were expressed as pico-gram/30 second and pico- gram/site in the 30-second GCF sample.

Amniotic membrane Lyophilized and irradiated AM (3×3 sq.cm) was obtained from a commercial tissue bank. The tissue was dispatched for clinical use from the tissue bank. The tissue conforms to the International Atomic Energy Agency (IAEA) recommendations and the Asia Pacific Association of Surgical Tissue Banks (APASTB) standards. AM is stable and can be stored at room temperature.

Surgical phase:

All surgical procedures were performed by one clinician. After recording relevant parameters, and following routine local anesthesia, sulcular incisions were given and full thickness mucoperiosteal flap was elevated for defect access. Thorough degranulation of the bone defect was done and root planing was done by using appropriate site-specific curettes.

The test site was treated as follows; After placement and proper condensation of natural Hydroxyapatite graft in the defect, AM was cut based on defect anatomy of surgical site and then adapted over the bone graft and alveolar bone extending from base of the flap reflection to the tooth surface. Flap was approximated and stabilized by placing direct loop sutures. Periodontal dressing was placed subsequently. For the control site, the procedure was identical except that the membrane was not placed. Patients received post-operative instructions and were prescribed medication. The sutures were removed at 1 week post-surgery and subsequent measures were recorded.

Radiographic assessment The evaluation of bone fill was performed by using digital subtraction technique and morphometric area analysis by using specific tools in two image processing softwares.

ELIGIBILITY:
Inclusion Criteria:

Systemically healthy chronic periodontitis patients within the age group of 30-55 years having at least 2 periodontal pockets ≥5 mm with at least 1 pocket in each quadrant showing radiographic evidence of vertical bone loss were included in the study. Assessment of suitability for GTR membrane placement was confirmed by transgingival probing to verify the presence of two well-contained interdental bone defects in as many quadrants.

Exclusion Criteria:

Smokers, medically compromised patients, pregnant women & lactating mothers and subjects receiving periodontal therapy in the 24 weeks (6-month)-period leading to the study were not included.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Actual)
Dates: Start 2012-03; Primary Completion 2013-02 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
The mean difference in levels of hBD-2/IL-1β | From Baseline to One month
  Commercially available ELISA kits were used to quantify GCF levels of hBD-2 and IL-1β. All assay procedures were conducted according to the manufacturer's instructions and in the test, 100μl of the samples or standards were added into the respective wells in duplicate. Color development was stopped using 1% H2SO4 and absorbance of the entire plate was measured within 30 minutes by an ELISA reader at 450nm. The amounts of hBD-2 and IL-1β were calculated based on the dilutions, and the results were expressed in picograms in the 30-second GCF sample.

SECONDARY OUTCOMES:
Bone fill assessment | Baseline to 6 months
  The evaluation of bone fill was performed by using digital subtraction technique and morphometric area analysis by using specific tools in two image processing software.

OTHER OUTCOMES:
Measures of periodontitis and gingivitis | Baseline to 6 months
  Non-invasive site-specific measures of the plaque index (PI) and modified gingival index (MGI) at the baseline, 1 week, 12 weeks and 24 weeks. The PPD, CAL and bone fill were recorded at the baseline (on the day of surgery) and at the end of 12 and 24 weeks. PPD and CAL were recorded at the baseline and at the end of 12 and 24 weeks using a UNC-15 color-coded periodontal probe.

CONTACTS AND LOCATIONS:
Overall Officials: Anumala Naveen, MDS, Study Chair — SVS Institute of Dental Sciences
Locations (1):
- SVS Institute of Dental Sciences, Mahabubnagar, Hyderabad, Andhra Pradesh, India